CLINICAL TRIAL: NCT06714318
Title: SMARTER: Using Blood Samples to iMprove FIT-bAsed coloRecTal cancEr scReening
Status: Recruiting | Type: Observational
Sponsor: Vejle Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: SMARTER
Record Dates: First submitted 2024-11-27; First posted 2024-12-03 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Screening participants: All citizens referred to colonoscopy at Vejle Hospital or Hospital Sønderjylland in the colorectal cancer screening program are offered to participate in the study. If the participant agrees, they will have blood drawn and sign a declaration of consent before their colonoscopy.

SUMMARY:
The project aims to investigate whether colorectal cancer screening can be improved using blood tests, thereby reducing the number of unnecessary colonoscopies. The Danish colorectal cancer screening program was implemented in 2014, and currently, all individuals aged 50-74 are invited every two years to participate. Those who test positive for hidden blood in their stool are referred for a colonoscopy. More than a third of the approximately 25,000 colonoscopies performed annually in the screening program can be classified as unnecessary, as they reveal a normal colon. This results in avoidable and unpleasant procedures for individuals and strains healthcare resources.

The project seeks to reduce the number of these unnecessary colonoscopies by investigating whether blood biomarkers can identify individuals at very low risk of colorectal cancer after a positive stool test for hidden blood. By utilizing blood tests, screening could become more personalized, precise, and resource-efficient for the healthcare system.

ELIGIBILITY:
Inclusion Criteria:

* Participation in the colorectal cancer screening program.

Exclusion Criteria:

* Participants are excluded if a colonoscopy is not completed unless this is due to a colorectal cancer obstruction.

Ages: 50 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All citizens referred to a colonoscopy at Vejle Hospital or Hospital Sønderjylland in the colorectal cancer screening program.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-12-02 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Correlation between result of blood test and colonoscopy result in patients screened positive for blood in the stool | From enrollment in study till 120 days after colonoscopy. The blood sample will be drawn before the colonoscopy and the final diagnosis from the colonoscopy will be registered 120 days after the colonoscopy.
  The aim is to investigate the individual's chance of being healthy despite a positive test for blood in the stool in the colorectal cancer screening program. The chance of being healthy is estimated from the combined blood sample results and will be compared to the results of the colonoscopy.

CONTACTS AND LOCATIONS:
Overall Officials: Jonna Skov Madsen, Prof., MD, Study Chair — Biochemistry and Immunology, Lillebaelt Hospital
Locations (2):
- Denmark (2):
  - Hospital Sønderjylland, Aabenraa
  - Vejle Hospital, Vejle

IPD SHARING:
Plan to Share IPD: Undecided